CLINICAL TRIAL: NCT04942873
Title: Study of Compliance and Influencing Factors in Chinese Patients With Nonvalvular Atrial Fibrillation (NVAF) to Oral Anticoagulant
Brief Title: The Adherence to Oral Anticoagulant in Chinese Patients With NVAF
Acronym: NVAF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-966
Record Dates: First submitted 2021-06-10; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Nonvalvular Atrial Fibrillation
Keywords: adherence; new oral anticoagulants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- dabigatran group: NVAF patients who taking dabigatran capsule 110mg，bid during 2016.2-2021.1，the duration of continuous medication was more than 3 months.PDC value and MMAS-8 scale were used to evaluate the compliance of patients with dabigatran.
  Interventions: Other: adherence
- Rivaroxaban group: NVAF patients who taking rivaroxaban tablet 15mg，bid during 2016.2-2021.1，the duration of continuous medication was more than 3 months.PDC value and mmas-8 scale were used to evaluate the compliance of patients with dabigatran. PDC value and mmas-8 scale were used to evaluate the compliance of patients with rivaroxaban.
  Interventions: Other: adherence
- wafarin group: NVAF patients who taking wafarin tablet during 2016.2-2021.1，the duration of continuous medication was more than 3 months， the dosage is adjusted according to INR. MMAS-8 scale was used to evaluate the compliance of patients with rivaroxaban.evaluate the compliance of patients with wafarin.
  Interventions: Other: adherence

INTERVENTIONS:
Other: adherence — PDC value and MMAS-8 scale were used to evaluate the compliance of patients with dabigatran, rivaroxaban and wafarin

SUMMARY:
Investigate the compliance of oral anticoagulants in Chinese NVAF patients and find out the causes, so as to provide basis for formulating effective measures to improve the compliance of oral anticoagulants.

DETAILED DESCRIPTION:
1. The general information about these patients was recorded such as gender, age, smoking history, drinking history, heart failure, hypertension, diabetes, coronary heart disease, stroke history, TIA history, peripheral vascular disease, etc. CHA2DS2-VASc score and HAS-BLED score were recorded.
2. Medication information and follow-up information was collected.For the patients included in the study, the medication records of oral anticoagulants (outpatient, emergency, hospitalization), adverse reactions, anticoagulant use history, drug withdrawal or dressing change, disease changes, etc. within three years were recorded by referring to the patient's medical records.

ELIGIBILITY:
Inclusion Criteria:

NVAF; CHA2DS2-VASc≥2（femal≥3）; After starting the medication, the duration of continuous medication was more than 3 months

Exclusion Criteria:

The patients had the records of anticoagulants in other hospitals; Patients lost to follow-up; Patients who do not need long-term anticoagulants after successful radiofrequency ablation or left atrial appendage occlusion. The follow-up time was 3 years or the following conditions occurred: the patient's condition changed and no longer used oral anticoagulants or died, the follow-up was stopped.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Through the hospital information system (HIS), the information of patients using warfarin, dabigatran and rivaroxaban during 2016.1-2-2021.1 was retrieved
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-07-20 (Estimated); Primary Completion 2022-06-06 (Estimated); Study Completion 2023-06-10 (Estimated)

PRIMARY OUTCOMES:
The long-term compliance of oral anticoagulants in NVAF patients was compared among warfarin group, dabigatran group and rivaroxaban group. | 6 months
  In this study, the eight item Morisky medication adherence scale (MMAS-8) was used to compare the long-term compliance of patients with warfarin, dabigatran axetil and rivaroxaban. The proportion of days covered (PDC) was used to compare the long-term compliance of patients with dabigatran and rivaroxaban.

SECONDARY OUTCOMES:
Explore the influence of different factors on patients' compliance, and to find out the factors influencing patients' long-term compliance, so as to provide basis for formulating strategies to improve patients' long-term compliance. | 6 months
  Data of all influencing factors included in CHA2DS2-VASc score scale, such as age hypertension，heart failure, diabetes, women and vascular diseases， as well as region, medical insurance category, education level, anticoagulant use history and HAS-BLED score
Through multivariate logistic regression analysis, to clarify the impact of various factors on long-term compliance of patients. | 6 months
  Univariate analysis of significant variables, further by multivariate logistic regression analysis

CONTACTS AND LOCATIONS:
Overall Officials: huang yuwen, master, Principal Investigator — The Second Affiliated Hospital of Medical College of Zhejiang University
Locations (1):
- Chang Cuie, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No